CLINICAL TRIAL: NCT00315172
Title: Non-Exercise Activity Thermogenesis (NEAT) in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060141; 06-CH-0141
Record Dates: First submitted 2006-04-15; First posted 2006-04-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-11-07

CONDITIONS: Non-exercise Activity Thermogenesis
Keywords: Adipose Tissue; Weight Gain; Pediatric; Body Composition; Thermogenesis; Exercise; Healthy Volunteer; HV
MeSH Terms: conditions — Weight Gain; Motor Activity

INTERVENTIONS:
Procedure: Non-Exercise Activity Thermogenesis (NEAT)

SUMMARY:
Non-exercise activity thermogenesis (NEAT) is the energy expended engaging in daily activities such as maintenance of posture, fidgeting, and other activities not specifically designated as "exercise." A growing body of evidence indicates that NEAT plays an important role in overall energy balance; for example, differences in NEAT account for the ease with which adults gain or lose weight during over- or under feeding. An intriguing and possibly modifiable component of NEAT is fidgeting-like activity. In lean and overweight adults, modulation of NEAT by augmenting fidgeting can increase short-term energy expenditure. It is unknown whether NEAT can be altered in children, or whether augmenting NEAT in children can change daily energy expenditure or body composition long-term. Children exhibit higher levels of daily activity than adults, suggesting potentially profound differences in energy balance. We propose to study the role of NEAT in children to determine if: a) the fidgeting component of NEAT can be measured accurately and reproducibly in children; b) NEAT can be increased by devices that remind children to engage in fidgeting-like activities; and c) manipulation of fidgeting-NEAT can significantly change energy expenditure and body composition. Thirty lean and thirty overweight children will be enrolled and treated in a pilot feasibility study. By adapting technologies developed to measure activity in adults, children's behavior and thermogenesis will be recorded and analyzed to study question (a). To address study questions (b) and (c), we will ask children to wear a timer that vibrate on a fixed interval schedule and be randomly assigned to two conditions: the intervention or active condition, during which children will be cued by the timer to engage in a fidgeting behavior (rapidly moving their heel up and down), and the control condition, during which children will be asked to perform a less thermogenic activity (noting the cue). Children will then cross over so that each child will complete both conditions. Primary outcome measures for question (a) will be changes in energy expenditure when subjects are asked to fidget in a laboratory environment. The correlation of these energy expenditure measurements with new activity monitoring technologies will also be obtained, so that such equipment can be used for measurements under free-living conditions. For study questions (b) and (c), compliance with prescribed fidgeting regimens in a free living environment and the changes in energy expenditure and body composition will be determined over a 2 week interval. This pilot study will enable the determination of the sample size needed to assess the efficacy of a longer term NEAT intervention in children.

DETAILED DESCRIPTION:
Non-exercise activity thermogenesis (NEAT) is the energy expended engaging in daily activities such as maintenance of posture, fidgeting, and other activities not specifically designated as "exercise." A growing body of evidence indicates that NEAT plays an important role in overall energy balance; for example, differences in NEAT account for the ease with which adults gain or lose weight during over- or under feeding. An intriguing and possibly modifiable component of NEAT is fidgeting-like activity. In lean and overweight adults, modulation of NEAT by augmenting fidgeting can increase short-term energy expenditure. It is unknown whether NEAT can be altered in children, or whether augmenting NEAT in children can change daily energy expenditure or body composition long-term. Children exhibit higher levels of daily activity than adults, suggesting potentially profound differences in energy balance. We propose to study the role of NEAT in children to determine if: a) the fidgeting component of NEAT can be measured accurately and reproducibly in children; b) NEAT can be increased by devices that remind children to engage in fidgeting-like activities; and c) manipulation of fidgeting-NEAT can significantly change energy expenditure and body composition. Thirty lean and thirty overweight children will be enrolled and treated in a pilot feasibility study. By adapting technologies developed to measure activity in adults, children's behavior and thermogenesis will be recorded and analyzed to study question (a). To address study questions (b) and (c), we will ask children to wear a timer that vibrate on a fixed interval schedule and be randomly assigned to two conditions: the intervention or active condition, during which children will be cued by the timer to engage in a fidgeting behavior (rapidly moving their heel up and down), and the control condition, during which children will be asked to perform a less thermogenic activity (noting the cue). Children will then cross over so that each child will complete both conditions. Primary outcome measures for question (a) will be changes in energy expenditure when subjects are asked to fidget in a laboratory environment. The correlation of these energy expenditure measurements with new activity monitoring technologies will also be obtained, so that such equipment can be used for measurements under free-living conditions. For study questions (b) and (c), compliance with prescribed fidgeting regimens in a free living environment and the changes in energy expenditure and body composition will be determined over a 2 week interval. This pilot study will enable the determination of the sample size needed to assess the efficacy of a longer term NEAT intervention in children.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria:

1. Good general health. Individuals taking medications for any serious medical condition will be excluded.
2. Age 7 to 11 years.
3. Body Mass Index 15th to 85th percentile for lean children or greater than or equal to 95% for age for overweight children.
4. Pre-pubertal (breast Tanner I - III for girls, testes size less than or equal to 10 mL for boys).

EXCLUSION CRITERIA:

Volunteers will be excluded for the following reasons:

1. Presence of major illnesses: renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing syndrome, untreated hyper- or hypothyroidism), hematological problems or pulmonary disorders.
2. Taking any medications that might interfere with weight or growth such as oral steroids, or psychotropic agents.
3. Presence of movement or tic disorders, since conditions increasing involuntary movements may interfere with the measurement of NEAT.
4. Individuals who are taking and/or have taken stimulant or weight loss medications in the last 6 months.
5. Individuals who cannot commit to living in a similar environment with similar levels of activity during the two weeks they wear the activity monitors and timer (i.e. cannot have one week wearing the activity monitors in school and the other week wearing the activity monitors on a ski vacation).
6. Intentional weight loss of more than 3 percent of body weight in the past two months.
7. Weight in excess of 300 lbs, because of the weight limits of the dual energy x-ray absorptiometry (DXA) scanners available at the NIH Clinical Center.
8. Inability to undergo MRI (e.g., volunteers with metal within their bodies including cardiac pacemakers, neural pacemakers, aneurysmal clips, shrapnel, ocular foreign bodies, cochlear implants, non-detachable electronic or electromechanical devices such as infusion pumps, nerve stimulators, bone growth stimulators, etc. that are contraindications).
9. Inability to tolerate study procedures at the screening visit.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Start 2006-04-13; Study Completion 2008-11-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Sorof JM, Lai D, Turner J, Poffenbarger T, Portman RJ. Overweight, ethnicity, and the prevalence of hypertension in school-aged children. Pediatrics. 2004 Mar;113(3 Pt 1):475-82. doi: 10.1542/peds.113.3.475. PMID 14993537
- [Derived] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099